CLINICAL TRIAL: NCT01817374
Title: A Pilot Study Evaluating Quantitative Volume Contrast Enhanced Ultrasound (VCEUS) Imaging for Determining Early Breast Cancer Response to Neoadjuvant Chemotherapy
Brief Title: Breast VCEUS to Evaluate Early Response to Neoadjuvant Chemotherapy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Principal Investigator, Mark E. Lockhart, Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: R12-021; 115,576 (Other: fda)
Record Dates: First submitted 2013-03-07; First posted 2013-03-25 (Estimated); Results first posted 2017-11-21 (Actual); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Definity; Ultrasound
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 2D US grayscale plus quantitative VCEUS (Other): Patients with breast cancer receiving neoadjuvant chemotherapy will undergo a 2D grayscale imaging followed by quantitative VCEUS imaging:
  1. prior to initiation of treatment (baseline);
  2. at 14 (± 4 days) after initiation of neoadjuvant chemotherapy (early treatment);
  3. at 28 days (± 4 days) after initiation of neoadjuvant chemotherapy (inter-regimen);
  4. at completion of therapy prior to definitive surgery (usually 2-3 months after initiation of treatment). Each patient will undergo a total of four VCEUS examinations.
  Interventions: Diagnostic Test: 2D US grayscale plus quantitative VCEUS

INTERVENTIONS:
Diagnostic Test: 2D US grayscale plus quantitative VCEUS — This is a pilot study to evaluate quantitative VCEUS imaging for determining early breast cancer response to neoadjuvant chemotherapy, comparing results with volume change on grayscale US and planar CEUS, and correlating imaging findings with pathological response on surgical specimens.
  Other Names: Definity VCEUS

SUMMARY:
1. Evaluate quantitative VCEUS imaging for determining early breast cancer response to neoadjuvant chemotherapy and compare results to co-temporal volume change on grayscale ultrasound and post-treatment mammography findings utilizing final surgical pathology and clinical outcome.
2. Assess incremental benefit of quantitative VCEUS to planar CEUS tumor perfusion measurements and enhancement patterns in predicting tumor response to adjuvant treatment in clinical studies.

The contrast agent Definity® is FDA approved for use as a contrast agent during ultrasound (echocardiography) of the heart. Definity® will be used "off-label" (during ultrasound of the breast) in this study. The administration of Definity® during this study will follow total dose guidelines approved by the FDA.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (age 19 years or older).
2. Patients with newly diagnosed and untreated stage II and III breast cancer scheduled to undergo neoadjuvant chemotherapy.
3. Patients with signed informed consent.

Exclusion Criteria:

1. Any history of prior radiation or chemotherapy for breast cancer.
2. Patients who only have non-measurable disease.
3. Patients who are medically unstable.
4. Patients with other primary cancers requiring systemic treatment.
5. Patients with cardiac shunts.
6. Patients with unstable cardiopulmonary conditions.
7. Patients with known pulmonary hypertension.
8. Patients with known hypersensitivity to any component of Definity (R) microbubble contrast.
9. Patients who are pregnant, breast-feeding or are planning to become pregnant during the study duration.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-06; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark E Lockhart, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 22 patients was planned in this pilot study through the UAB Interdisciplinary Breast Center. However, due to early termination of the study, only six breast cancer patients were enrolled. Each participant received both interventions (2D ultrasound grayscale vs Definity Volume contrast enhanced ultrasound).
Pre-assignment Details: Recruitment for this study started in June 2015. The primary completion point was reached at July 2016, and study completion July 2016. The study was conducted at the University of Alabama at Birmingham.
Groups:
- Evaluation of VCEUS to Determine Response to Chemotherapy: Patients with breast cancer receiving neoadjuvant chemotherapy will undergo 2D grayscale imaging followed by the quantitative VCEUS imaging as follows:
  1. prior to initiation of treatment (baseline);
  2. at 14 (± 4 days) after initiation of neoadjuvant chemotherapy (early treatment);
  3. at 28 days (± 4 days) after initiation of neoadjuvant chemotherapy (inter-regimen);
  4. at completion of therapy prior to definitive surgery (usually 2-3 months after initiation of treatment). Each patient will undergo a total of four VCEUS examinations.
  Definity (Perflutren Lipid Microspheres): This is a pilot study to evaluate quantitative VCEUS imaging for determining early breast cancer response to neoadjuvant chemotherapy, comparing results with volume change on grayscale US and planar CEUS, and correlating imaging findings with pathological response on surgical specimens.
Period: Overall Study
Arm/Group | Evaluation of VCEUS to Determine Response to Chemotherapy
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Total number of participants is 6. All participants received both interventions.
Groups:
- Evaluation of VCEUS to Determine Response to Chemotherapy: Patients with breast cancer receiving neoadjuvant chemotherapy will undergo quantitative VCEUS imaging and 2D grayscale imaging as follows:
  1. prior to initiation of treatment (baseline);
  2. at 14 (± 4 days) after initiation of neoadjuvant chemotherapy (early treatment);
  3. at 28 days (± 4 days) after initiation of neoadjuvant chemotherapy (inter-regimen);
  4. at completion of therapy prior to definitive surgery (usually 2-3 months after initiation of treatment). Each patient will undergo a total of four VCEUS examinations.
  Definity (Perflutren Lipid Microspheres): This is a pilot study to evaluate quantitative VCEUS imaging for determining early breast cancer response to neoadjuvant chemotherapy, comparing results with volume change on grayscale US and planar CEUS, and correlating imaging findings with pathological response on surgical specimens.
Arm/Group | Evaluation of VCEUS to Determine Response to Chemotherapy
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Tumor Volume Measure Using Grayscale US
Description: Grayscale ultrasound (standard of care) size in millimeters along the longest axis. Range of the grayscale is a minimum of 21.0 millimeters and maximum of 82 millimeters.
Time Frame: Baseline (first visit)
Measure: Mean (Standard Deviation); unit: millimeters
Groups:
- Grayscale Ultrasound: Patients with breast cancer receiving neoadjuvant chemotherapy will undergo a 2D grayscale imaging prior to initiation of treatment (baseline);
Arm/Group | Grayscale Ultrasound
Number analyzed (Participants) | 6
millimeters | 38.2 (23.9)

2. Primary Outcome: VCEUS Perfusion Time to Peak
Description: Time of maximal perfusion relative to contrast injection. Range for time to peak intensity is a minimum of 67.5 seconds and a maximum of 99.0 seconds.
Time Frame: Baseline
Population: 1 subject did not complete this timepoint due to machine down
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- VCEUS Perfusion Time to Peak: Time from contrast injection to peak intensity
Arm/Group | VCEUS Perfusion Time to Peak
Number analyzed (Participants) | 5
seconds | 88.5 (12.9)

3. Primary Outcome: Tumor Volume Measure Using Grayscale US
Description: as for outcome 1
Time Frame: Week 2
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Grayscale Ultrasound
Number analyzed (Participants) | 6
millimeters | 34.0 (29.9)

4. Primary Outcome: Tumor Volume Measure Using Grayscale US
Description: as for outcome 1
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Grayscale Ultrasound
Number analyzed (Participants) | 6
millimeters | 27.3 (22.4)

5. Primary Outcome: Tumor Volume Measure Using Grayscale US
Description: as for outcome 1
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Grayscale Ultrasound
Number analyzed (Participants) | 6
millimeters | 18.0 (9.01)

6. Primary Outcome: VCEUS Perfusion Time to Peak
Description: as for outcome 2
Time Frame: Week 2
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | VCEUS Perfusion Time to Peak
Number analyzed (Participants) | 6
seconds | 85.7 (24.4)

7. Primary Outcome: VCEUS Perfusion Time to Peak
Description: as for outcome 2
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | VCEUS Perfusion Time to Peak
Number analyzed (Participants) | 6
seconds | 88.3 (29.8)

8. Primary Outcome: VCEUS Perfusion Time to Peak
Description: as for outcome 2
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | VCEUS Perfusion Time to Peak
Number analyzed (Participants) | 6
seconds | 105.16 (43.2)

9. Secondary Outcome: Pathology Residual Tumor
Description: Pathology residual tumor measured in millimeters
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: millimeters
Groups:
- Pathology Residual: Pathology residual tumor measured in millimeters
Arm/Group | Pathology Residual
Number analyzed (Participants) | 6
millimeters | 34.5 (28.8)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from Baseline through 3 months..
Groups:
- Definity VCEUS: Patients with breast cancer receiving neoadjuvant chemotherapy will undergo quantitative VCEUS imaging and 2D grayscale imaging as follows:
  1. prior to initiation of treatment (baseline);
  2. at 14 (± 4 days) after initiation of neoadjuvant chemotherapy (early treatment);
  3. at 28 days (± 4 days) after initiation of neoadjuvant chemotherapy (inter-regimen);
  4. at completion of therapy prior to definitive surgery (usually 2-3 months after initiation of treatment). Each patient will undergo a total of four VCEUS examinations.
  Definity (Perflutren Lipid Microspheres): This is a pilot study to evaluate quantitative VCEUS imaging for determining early breast cancer response to neoadjuvant chemotherapy, comparing results with volume change on grayscale US and planar CEUS, and correlating imaging findings with pathological response on surgical specimens.
Arm/Group | Definity VCEUS
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No